CLINICAL TRIAL: NCT07280039
Title: Mortality and Muscle Mass Loss in Critically Ill Patients: A Prospective, Observational, Multicenter Study.
Brief Title: Mortality and Muscle Mass Loss in Critically Ill Patients.
Acronym: MUSIC 2
Status: Not yet recruiting | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Roman Gal, head of the department, Brno University Hospital
Other Study IDs: CT0022025
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Mortality; Muscle Loss
Keywords: Mortality; Muscle loss; Muscle ultrasound; Critically ill; Rectus femoris cross area
MeSH Terms: conditions — Muscular Atrophy; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to monitor changes in muscle mass in critically ill patients and to verify whether a decrease in muscle mass of ≥10% during the first 7 days of hospitalization is associated with increased 28-day mortality. We will be used ultrasoud for measurement the rectus femoris cross sectional area.

DETAILED DESCRIPTION:
All patients will be admitted to participating ICU centers from December 2025 to December 2026 will be screened and enrolled based on the inclusion and exclusion criteria. Informed consent will be requested. Ultrasound measurements will be performed by the same investigator within the first 24h after ICU admssion and again on day 7 of the patient´s ICU stay. All patient data will be entered into case report form by a study physician. In the follow-up will be determined 28 mortality.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* mechanical ventilation expected for at least 48 hours

Exclusion Criteria:

* Clinical Frailty Score above 7 prior admission
* Neuromuscular disease in previous medical history
* Amputated lower extremities
* Trauma of lower extremities involving tights
* Conditions affecting the nervous system with involvement of the thigh muscle
* Inability to cooperate during ultrasound examination
* Inability to perform ultrasound examination on day 7

  9. Inability to perform ultrasound examination on day 7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients will be admitted to intensive care unit with suspect length of artificial ventilation more than 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Relationship between muscle loss and 28 day mortality | 28 days after enrollment
  Critically ill patients with a ≥10% decrease in rectus femoris cross-sectional area have increased 28 day mortality.

SECONDARY OUTCOMES:
Incidence of a significant decrease in rectus femoris cross-sectional area | first 7 days of ICU stay
  A decrease in rectus femoris cross-sectional area of 10% or more measured by ultrasound.
Incidence of an insignificant decrease in rectus femoris cross-sectional area | first 7 days ICU stay
  A decrease in rectus femoris cross-sectional area of less than 10% measured by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gal, M.D., PhD, Study Chair — The University Hospital Brno
Locations (1):
- The University Hospital Brno, Brno, Bohunice, Czechia

IPD SHARING:
Plan to Share IPD: No